CLINICAL TRIAL: NCT05487053
Title: The Impact of Single-shot Adductor Canal Block Versus Continuous Femoral Nerve Block on Rehabilitation After Total Knee Replacement (AdORe - ACB)
Brief Title: The Impact of Single-shot Adductor Canal Block Versus Continuous Femoral Nerve Block on Rehabilitation After Total Knee Replacement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Negovsky Reanimatology Research Institute (Other Government)
Responsible Party: Principal Investigator, Valery Likhvantsev, MD, Head of the Research V. Negovsky Reanimatology Research Institute, Negovsky Reanimatology Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AdORe - ACB
Record Dates: First submitted 2022-08-03; First posted 2022-08-04 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Osteo Arthritis Knee; Gonarthrosis
Keywords: Osteo Arthritis Knee; Gonarthrosis; Regional anesthesia; Analgesia; Postoperative analgesia; Total knee replacement; Continuous femoral nerve block; Femoral nerve block; Continuous adductor canal block; Adductor canal block
MeSH Terms: conditions — Osteoarthritis, Knee; Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single-shot adductor canal block (Experimental)
  Interventions: Procedure: Single-shot adductor canal block
- Continuous femoral nerve block (Active Comparator)
  Interventions: Procedure: Continuous femoral nerve block

INTERVENTIONS:
Procedure: Single-shot adductor canal block — Postoperative analgesia in this group will be carried out by a single-shot bolus of 20 ml Ropivacaine 0.5% in the region of the middle third of the adductor canal.
  Arms: Single-shot adductor canal block
Procedure: Continuous femoral nerve block — Postoperative analgesia in this group will be carried out by continuous infusion of local anesthetics through a catheter installed to the femoral nerve in the area of the femoral triangle. Ropivacaine 0.2% solution will be used for postoperative analgesia. Local anesthetic infusion rate is 4 ml/h to 10 ml/h.
  Arms: Continuous femoral nerve block

SUMMARY:
Total knee replacement (TKR) is considered the most effective and safe method of radical treatment of late stages of knee osteoarthritis. A well-known problem of TKR is a severe postoperative pain syndrome, which is observed in more than 50% of patients.

Femoral nerve block (FNB) is the "gold standard" for continuous postoperative analgesia after total knee replacement, as it is effective in reducing the frequency of use of opioid analgetics and reduce the duration of hospitalization. At the same time, the negative effect of this method is the motor blockade of the quadriceps femoris muscle which leads to functional impairment and is associated with an increased risk of falling.

Adductor canal block (ACB) provides adequate analgesia comparable to femoral nerve block. Moreover, ACB doesn't affect the motor function of the quadriceps femoris muscle.

The possibility of enhanced recovery after total knee replacement is the reason to compare single-shot adductor canal block and continuous femoral nerve block.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Planned primary total knee replacement
* Planned neuraxial anesthesia
* Written informed consent

Exclusion Criteria:

* Urgent surgery
* Planned revision total knee replacement
* Known allergic reaction to anesthetics
* Confirmed localized infection at the puncture sites
* Confirmed localized tumor at the puncture sites
* Peripheral neuropathy of the lower extremities
* Parkinson's disease
* Previously enrolled in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-02-03 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Ambulation distance | postoperative day 1
  Less meters means worse outcome

SECONDARY OUTCOMES:
Ambulation distance | postoperative day 2
  Less meters means worse outcome
Timed up and go test | postoperative day 1
  More seconds means worse outcome
Timed up and go test | postoperative day 2
  More seconds means worse outcome
10 meters walk test | postoperative day 1
  More seconds means worse outcome
10 meters walk test | postoperative day 2
  More seconds means worse outcome
30 seconds chair stand test | postoperative day 1
  Less exercise done means worse outcome
30 seconds chair stand test | postoperative day 2
  Less exercise done means worse outcome
5 times sit to stand test | postoperative day 1
  More seconds means worse outcome
5 times sit to stand test | postoperative day 2
  More seconds means worse outcome
time to readiness to dicharge | 30 day
  time from the day of surgery to the day of readiness to discharge
length of hospitalization | 30 day
  time from the day of surgery to the day of discharge

OTHER OUTCOMES:
intravascular local anesthetic injection | 30 day
  frequency of intravascular local anesthetic injection
neuropathy after the procedure | 30 day
  frequency of neuropathy after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Valery Likhvantsev, Principal Investigator — Negovsky Reanimatology Research Institute
Locations (1):
- Clinical Hospital on Yauza, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No